CLINICAL TRIAL: NCT04981366
Title: Effects of the Protein Supplementation Associated With Exercise Training in Elderly With Sarcopenic Obesity Undergoing Caloric Restriction
Brief Title: Protein Supplementation in Elderly With Sarcopenic Obesity Undergoing Caloric Restriction and Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Hamilton Augusto Roschel da Silva, Principal Investigator, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04234918.1.0000.0065
Record Dates: First submitted 2021-07-01; First posted 2021-07-29 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Sarcopenic Obesity; Aging

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (CTRL) (No Intervention): Patients allocated to this arm will not receive any intervention.
- Caloric Restriction associated to exercise training plus protein supplementation (CREX+PTN) (Experimental): Patients allocated to this arm will be submitted to caloric restriction associated with exercise training program plus protein supplementation.
  Interventions: Dietary Supplement: Protein supplement
- Caloric Restriction associated to exercise training plus isocaloric placebo (CREX+PLA) (Placebo Comparator): Patients allocated to this arm will be submitted to caloric restriction associated with exercise training program plus isocaloric placebo.
  Interventions: Dietary Supplement: isocaloric supplement

INTERVENTIONS:
Dietary Supplement: Protein supplement — 40g of whey protein in the breakfast;
  Arms: Caloric Restriction associated to exercise training plus protein supplementation (CREX+PTN)
Dietary Supplement: isocaloric supplement — 42g of isocaloric supplement in the breakfast;
  Arms: Caloric Restriction associated to exercise training plus isocaloric placebo (CREX+PLA)

SUMMARY:
This study aims to investigate if protein supplementation increases the benefits of exercise training in the elderly with sarcopenic obesity undergoing caloric restriction.

DETAILED DESCRIPTION:
A major subset of adults over the age of 65 is now classified as having sarcopenic obesity, a high-risk geriatric syndrome predominantly observed in an aging population that is at risk of synergistic complications from both sarcopenia and obesity.

Lifestyle interventions such as caloric restriction and exercise training are effective nonpharmacological strategies to mitigate some adverse effects related to this condition. Also, protein supplementation may boost the benefits of exercise, but this assumption is still to be tested. This trial aims to test whether protein supplementation is able to increase the benefits of exercise training in the elderly with sarcopenic obesity undergoing caloric restriction.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and older;
* Body mass index (BMI) > 30 kg/m2;
* Sarcopenia;
* not engage into exercise training programas.

Exclusion Criteria:

* cancer in the last 5 years;
* cognitive deficit or dementia that impossibility the patient to read and sign the informed consent form;
* any disease that limits participation in exercise training program.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hamilton Roschel, Phd, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started: 2021-08-01 Recruitment finished: 2023-02-26
Groups:
- Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN): Patients allocated to this arm were submitted to caloric restriction associated with an exercise training program plus protein supplementation.
  Protein supplement: 40g of whey protein in the breakfast;
- Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA): Patients allocated to this arm were submitted to caloric restriction associated with an exercise training program plus isocaloric placebo.
  isocaloric supplement: 42g of non-nitrogenous, isocaloric supplement in the breakfast;
- Control Group (CTRL): Patients allocated to this arm did not receive any intervention.
Period: Overall Study
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Started | 35 | 35 | 35
Completed | 29 | 29 | 27
Not Completed | 6 | 6 | 8
Not completed — Withdrawal by Subject | 5 | 4 | 8
Not completed — Health issues unrelated to the trial | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL) | Total
Number analyzed (Participants) | 35 | 35 | 35 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] — Participant age was recorded in years at the time of study enrollment
  years | 72.2 (5.6) | 71.8 (5.6) | 71.1 (5.3) | 71.7 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 27 | 27 | 81
  Male | 8 | 8 | 8 | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Brazil | 35 | 35 | 35 | 105
Body mass index (kg/m²) [Mean (Standard Deviation); unit: kg/m²] — Body mass index was calculated by dividing the body weight by squared height.
  kg/m² | 36.0 (4.8) | 34.8 (4.5) | 34.5 (4) | 35.1 (4.4)
Total fat-free mass (%) [Mean (Standard Deviation); unit: Percentage] — Total fat-free mass was evaluated using the dual X-ray absorptiometry
  Percentage | 49.6 (5.4) | 50.3 (4.8) | 50.5 (5.1) | 50.2 (5.1)
Appendicular fat-free mass (kg) [Mean (Standard Deviation); unit: Kg] — Appendicular fat-free mass was evaluated using dual X-ray absorptiometry and was considered as the sum of fat-free mass of upper and lower limbs.
  Kg | 17.7 (4.2) | 18.0 (3.7) | 17.4 (3.6) | 17.7 (3.8)
Appendicular fat-free mass to body mass index ratio [Mean (Standard Deviation); unit: Kg/Kg/m^2] — Appendicular fat-free mass/BMI was calculated as the ratio of appendicular fat-free mass to body mass index.
  Kg/Kg/m^2 | 0.49 (0.12) | 0.52 (0.11) | 0.51 (0.10) | 0.51 (0.11)
Leg fat-free mass (kg) [Mean (Standard Deviation); unit: Kg] — Leg fat-free mass was evaluated using dual X-ray absorptiometry and was considered as the sum of the fat-free mass of lower limbs.
  Kg | 13.5 (3.2) | 13.5 (2.7) | 13.2 (2.7) | 13.4 (2.9)
Diabetes (n) [Count of Participants; unit: Participants] | 11 | 12 | 7 | 30
Hypertension (n) [Count of Participants; unit: Participants] | 29 | 20 | 23 | 72
Psychiatric diseases (n) [Count of Participants; unit: Participants] | 6 | 12 | 5 | 23
Rheumatic diseases (n) [Count of Participants; unit: Participants] | 4 | 3 | 6 | 13
Dyslipidemia (n) [Count of Participants; unit: Participants] | 16 | 15 | 13 | 44
Osteopenia (n) [Count of Participants; unit: Participants] | 21 | 20 | 21 | 62

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Fat-free Mass
Description: Fat-free mass evaluated through dual-energy x-ray absorptiometry (DEXA) and reported as percentage
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: percentage of fat-free mass
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
percentage of fat-free mass
  Pre | 49.6 (5.4) | 50.3 (4.8) | 50.5 (5.1)
  Post | 52.5 (5.9) | 52.7 (4.3) | 49.3 (4.7)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.013, Mixed Models Analysis — We applied the restricted maximum likelihood, compound symmetry covariance structure, and Kenward-Roger degrees of freedom approximation. To maintain the significance level at 0.05, the primary endpoints were assessed using Hochberg's procedure

2. Primary Outcome: Appendicular Fat-free Mass
Description: Appendicular fat-free mass was evaluated through dual-energy x-ray absorptiometry (DEXA) and calculated as the sum of the fat-free mass of the upper and lower limbs.
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
Kg
  Pre | 17.7 (4.2) | 18.0 (3.7) | 17.4 (3.6)
  Post | 18.1 (3.5) | 17.6 (3.5) | 16.5 (2.7)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

3. Primary Outcome: Appendicular Fat-free Mass to Body Mass Index Ratio
Description: The appendicular fat-free mass (AFFM) was assessed using dual-energy X-ray absorptiometry (DXA) and expressed in kilograms (kg). The body mass index (BMI) was calculated as weight in kilograms divided by the square of height in meters (kg/m²). The AFFM/BMI ratio was computed by dividing AFFM (kg) by BMI (kg/m²), resulting in a unitless ratio. Higher values indicate greater muscle mass relative to body size
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: Kg/Kg/m^2
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
Kg/Kg/m^2
  Pre | 0.49 (0.12) | 0.52 (0.11) | 0.51 (0.10)
  Post | 0.54 (0.11) | 0.54 (0.11) | 0.48 (0.09)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p < 0.001, Mixed Models Analysis

4. Primary Outcome: Leg Fat-free Mass
Description: Appendicular fat-free mass was evaluated through dual-energy x-ray absorptiometry (DEXA) and calculated as the sum of the fat-free mass of the lower limbs.
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
Kg
  Pre | 13.5 (3.2) | 13.5 (2.7) | 13.2 (2.7)
  Post | 13.8 (2.6) | 13.0 (2.5) | 12.5 (2.2)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.007, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

5. Secondary Outcome: Fat-mass
Description: Fat mass was evaluated trough dual-energy x-ray absorptiometry (DEXA) and reported as percentage.
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: percentage of fat mass
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
percentage of fat mass
  Pre | 48.6 (5.6) | 47.8 (4.9) | 47.7 (5.2)
  Post | 45.6 (6.0) | 45.4 (4.4) | 48.9 (4.9)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p < 0.001, Mixed Models Analysis

6. Secondary Outcome: Quadriceps Cross-sectional Area (CSA)
Description: Quadriceps cross-sectional area (CSA) was assessed by computed tomography imaging
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: cm²
Groups:
- Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA): Patients allocated to this arm were submitted to caloric restriction associated with an exercise training program plus isocaloric placebo.
  socaloric supplement: 42g of non-nitrogenous, isocaloric supplement in the breakfast;
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
cm²
  Pre | 51.7 (13.4) | 50.7 (12.1) | 50.1 (14.4)
  Post | 54.3 (13.4) | 51.9 (12.9) | 47.7 (11.5)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p < 0.001, Mixed Models Analysis

7. Secondary Outcome: Rectus Femoris Cross-sectional Area (CSA)
Description: Rectus femoris cross-sectional area (CSA) was assessed by B-mode ultrasound.
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: cm²
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
cm²
  Pre | 3.39 (1.06) | 3.23 (0.96) | 3.32 (1.21)
  Post | 3.45 (1.07) | 3.27 (0.95) | 3.10 (0.98)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.005, Mixed Models Analysis

8. Secondary Outcome: Vastus Lateralis Cross-sectional Area (CSA)
Description: Vastus lateralis cross-sectional area (CSA) was assessed by B-mode ultrasound.
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: cm²
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
cm²
  Pre | 12.32 (2.69) | 12.15 (2.84) | 12.13 (3.53)
  Post | 12.55 (2.84) | 12.45 (2.77) | 11.49 (2.81)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p < 0.001, Mixed Models Analysis

9. Secondary Outcome: Muscle Fiber Cross-sectional Area (fCSA)- Type I
Description: Muscle fiber cross-sectional area (type I) was assessed using an immunostaining assay of muscle tissue samples obtained through percutaneous muscle biopsy
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Population: This exploratory subgroup analysis included only participants who consented to undergo a muscle biopsy (n = 20 out of 105 total participants).
Measure: Mean (Standard Deviation); unit: µm²
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 6 | 7 | 7
µm²
  Pre | 2240.7 (901.5) | 2725.8 (1121.6) | 2669.4 (806.7)
  Post | 3108.6 (1212.8) | 2859.4 (948.67) | 2614.6 (1076.4)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p < 0.001, Mixed Models Analysis

10. Secondary Outcome: Muscle Fiber Cross-sectional Area (fCSA)- Type II
Description: Muscle fiber cross-sectional area (type II) was assessed using an immunostaining assay of muscle tissue samples obtained through percutaneous muscle biopsy
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: µm²
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 6 | 7 | 7
µm²
  Pre | 2175.6 (827.6) | 2401.4 (1108.8) | 2340.8 (921.2)
  Post | 2775.2 (964.1) | 2239.5 (724.8) | 2166.1 (979.8)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p < 0.001, Mixed Models Analysis

11. Secondary Outcome: Serum Levels of C-terminal Telopeptide of Type I Collagen (CTX-I)
Description: Bone turnover was assessed by an automated electrochemiluminescence method.
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 29 | 29 | 27
ng/mL
  Pre | 0.34 (0.19) | 0.38 (0.18) | 0.35 (0.13)
  Post | 0.38 (0.22) | 0.46 (0.21) | 0.35 (0.12)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p < 0.001, Mixed Models Analysis

12. Secondary Outcome: Serum Levels of Procollagen Type I N-terminal Propeptide - (P1NP)
Description: Bone turnover was assessed by an automated electrochemiluminescence method.
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 29 | 29 | 27
ng/mL
  Pre | 53.1 (21.2) | 61.0 (26.9) | 56.3 (22.8)
  Post | 66.2 (61.0) | 66.1 (32.2) | 56.8 (22.7)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.001, Mixed Models Analysis

13. Secondary Outcome: Bone Mineral Density (Whole-body)
Description: bone mineral density (whole-body) evaluated trough dual-energy x-ray absorptiometry (DEXA)
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: g/cm²
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
g/cm²
  Pre | 1.08 (0.11) | 1.10 (0.11) | 1.05 (0.12)
  Post | 1.06 (0.11) | 1.08 (0.11) | 1.05 (0.11)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.033, Mixed Models Analysis

14. Secondary Outcome: Bone Mineral Density (Femur Neck)
Description: bone mineral density (femur neck) evaluated trough dual-energy x-ray absorptiometry (DEXA)
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: g/cm²
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
g/cm²
  Pre | 0.75 (0.11) | 0.75 (0.11) | 0.74 (0.11)
  Post | 0.74 (0.12) | 0.75 (0.12) | 0.74 (0.11)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.944, Mixed Models Analysis

15. Secondary Outcome: Bone Mineral Density (Total Hip)
Description: bone mineral density (total hip) evaluated trough dual-energy x-ray absorptiometry (DEXA)
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: g/cm²
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
g/cm²
  Pre | 0.90 (0.13) | 0.93 (0.11) | 0.89 (0.13)
  Post | 0.90 (0.13) | 0.93 (0.12) | 0.88 (0.13)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.203, Mixed Models Analysis

16. Secondary Outcome: Bone Mineral Density (Lumbar Spine)
Description: bone mineral density (lumbar spine) evaluated trough dual-energy x-ray absorptiometry (DEXA)
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: g/cm²
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
g/cm²
  Pre | 0.98 (0.12) | 1.01 (0.16) | 0.96 (0.15)
  Post | 0.97 (0.12) | 1.00 (0.16) | 0.96 (0.14)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.027, Mixed Models Analysis

17. Secondary Outcome: Bone Microarchitecture (Total Volumetric Density)
Description: Bone microarchitecture (total volumetric density) was assessed at the distal region of the radius of the non-dominant limb using a high-resolution peripheral quantitative computed tomography (HR-pQCT)
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: mg HA/cm³
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
mg HA/cm³
  Pre | 331.9 (82.0) | 309.5 (58.9) | 324.7 (75.4)
  Post | 340.2 (85.2) | 308.6 (66.8) | 328.9 (72.9)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.145, Mixed Models Analysis

18. Secondary Outcome: Bone Microarchitecture (Trabecular Volumetric Density)
Description: Bone microarchitecture (trabecular volumetric density) was assessed at the distal region of the radius of the non-dominant limb using a high-resolution peripheral quantitative computed tomography (HR-pQCT)
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: mg HA/cm³
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
mg HA/cm³
  Pre | 147.7 (37.8) | 309.5 (58.9) | 324.7 (75.4)
  Post | 152.0 (37.9) | 308.6 (66.8) | 328.9 (72.9)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.001, Mixed Models Analysis

19. Secondary Outcome: Bone Microarchitecture (Cortical Volumetric Density)
Description: Bone microarchitecture (cortical volumetric density) was assessed at the distal region of the radius of the non-dominant limb using a high-resolution peripheral quantitative computed tomography (HR-pQCT)
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: mg HA/cm³
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
mg HA/cm³
  Pre | 969.9 (59.8) | 951.0 (76.1) | 972.8 (60.3)
  Post | 969.9 (62.5) | 948.7 (76.3) | 975.5 (57.5)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.551, Mixed Models Analysis

20. Secondary Outcome: Bone Microarchitecture (BV/TV)
Description: Bone microarchitecture (BV/TV) was assessed at the distal region of the radius of the non-dominant limb using high-resolution peripheral quantitative computed tomography (HR-pQCT). Specifically, trabecular bone volume fraction (BV/TV) is computed as the ratio of the trabecular bone mineral density (Tb.vBMD in mg HA/cm3) and 1200 mg HA/cm3, which is assumed to be the density of fully mineralized bone. Afterwards, the values were multiplied by 100 to reflect the percentage of trabecular bone volume fraction.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: percentage of trabecular bone volume
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
percentage of trabecular bone volume
  Pre | 12.5 (3.2) | 12.9 (2.8) | 12.2 (3.0)
  Post | 12.7 (3.5) | 12.9 (3.0) | 12.3 (3.2)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.001, Mixed Models Analysis

21. Secondary Outcome: Bone Microarchitecture (Trabecular Number - Tb. N)
Description: The trabecular number (Tb.N) was analyzed using the ridge extraction technique in high-resolution peripheral quantitative computed tomography (HR-pQCT). In this approach, the trabeculae were treated as elongated structures resembling ridges. The technique involves detecting the central axis (ridge) of each trabecular element in a 3D image.
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: Trabeculae per mm
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
Trabeculae per mm
  Pre | 1.86 (0.35) | 1.96 (0.33) | 1.90 (0.38)
  Post | 1.90 (0.33) | 1.93 (0.34) | 1.90 (0.35)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.001, Mixed Models Analysis

22. Secondary Outcome: Bone Microarchitecture (Trabecular Separation)
Description: Trabecular separation (Tb.Sp), represents the average distance between trabeculae in the trabecular bone region. It was assessed using the distance transformation method, applied to the background (void space) of the trabecular structure. The transformation method measures the distance from each voxel (3D pixel) in the void space to the nearest trabecular element, and the average of these distances is then calculated. This method enables precise quantification of trabecular spacing in high-resolution 3D images.
  The separation is inversely related to trabecular density, as closer trabeculae indicate a higher bone volume fraction (BV/TV) and a denser bone network. The calculation of trabecular separation can be expressed as:
  Tb.Sp = 1- BV/TV : Tb.N
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
mm
  Pre | 0.493 (0.127) | 0.459 (0.092) | 0.488 (0.132)
  Post | 0.474 (0.101) | 0.474 (0.106) | 0.469 (0.117)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.001, Mixed Models Analysis

23. Secondary Outcome: Bone Microarchitecture (Trabecular Thickness)
Description: Trabecular thickness (Tb.Th) represents the average thickness of trabecular bone elements. It was assessed by calculating the mean thickness of the segmented trabecular structure, using the distance transformation method applied to the trabecular bone tissue.
  The trabecular thickness is calculated as a ratio of the bone volume fraction (BV/TV) to trabecular number (Tb.N): Tb.Th =BV/TV : Tb.N
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
mm
  Pre | 0.066 (0.014) | 0.066 (0.013) | 0.066 (0.012)
  Post | 0.064 (0.013) | 0.068 (0.012) | 0.067 (0.011)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.008, Mixed Models Analysis

24. Secondary Outcome: Bone Microarchitecture (Cortical Porosity)
Description: Cortical porosity (Ct.Po) is quantified using a density-based approach that segments bone into three compartments: compact cortex, transitional zone, and trabecular compartment. Voxels with a density below 1000 mg HA/cm³ indicate the presence of void space (pores), and porosity is estimated as the ratio of void space in each voxel. The mean of this ratio is calculated across all voxels in the compartment of interest, and the values were multiplied by 100. This method captures pores with diameters below the scanner's spatial resolution but relies on the assumption of fixed bone tissue mineral density and may be susceptible to image noise and beam hardening.
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
percentage
  Pre | 3.5 (2.5) | 3.5 (2.2) | 3.2 (2.4)
  Post | 3.1 (1.3) | 3.4 (2.6) | 3.5 (2.5)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p < 0.001, Mixed Models Analysis

25. Secondary Outcome: Bone Microarchitecture (Cortical Thickness)
Description: Bone microarchitecture (cortical thickness) wwas assessed at the distal region of the radius of the non-dominant limb using a high-resolution peripheral quantitative computed tomography (HR-pQCT)
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
mm
  Pre | 0.958 (0.242) | 0.827 (0.201) | 0.908 (0.193)
  Post | 0.968 (0.240) | 0.826 (0.203) | 0.911 (0.203)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.344, Mixed Models Analysis

26. Secondary Outcome: Bone Microarchitecture (Cortical Pore Diameter)
Description: Bone microarchitecture (cortical pore diameter) was assessed at the distal region of the radius of the non-dominant limb using a high-resolution peripheral quantitative computed tomography (HR-pQCT)
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
mm
  Pre | 0.168 (0.038) | 0.172 (0.043) | 0.169 (0.029)
  Post | 0.166 (0.038) | 0.174 (0.038) | 0.171 (0.030)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.613, Mixed Models Analysis

27. Secondary Outcome: Bone Microarchitecture (Stiffness)
Description: Stiffness (kN/mm) is defined as the total reaction force of the model divided by the applied displacement. It represents the resistance of a material or structure to deformation under an applied load. A higher stiffness value indicates greater resistance to deformation, while a lower value suggests more flexibility.
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: kN/mm
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
kN/mm
  Pre | 72.7 (20) | 74.1 (18.6) | 71.6 (20.2)
  Post | 73.5 (18.9) | 75.1 (19.6) | 69.7 (18.2)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.944, Mixed Models Analysis

28. Secondary Outcome: Bone Microarchitecture (Estimated Failure Load)
Description: Estimated failure load is indirectly calculated from linear finite element (FE) models using a yield criterion. The failure load is estimated when a specified volume of bone tissue (critical volume) exceeds a critical strain threshold, at which point the model is assumed to have yielded. This approach is often based on the Pistoia criterion, which is used to predict the point of failure in the material based on its mechanical properties and deformation behavior.
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: kN
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
kN
  Pre | 3458 (910) | 3553 (888) | 3430 (948)
  Post | 3503 (860) | 3598 (940) | 3347 (863)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.601, Mixed Models Analysis

29. Secondary Outcome: Isometric Muscle Strength - Handgrip
Description: Isometric muscle strength was evaluated using a handgrip dynamometer (Jamar®, Sammons Preston Rolyan, USA).
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
Kg
  Pre | 18.57 (5.44) | 19.29 (5.84) | 19.86 (5.62)
  Post | 23.17 (5.38) | 23.71 (4.82) | 18.43 (5.07)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p < 0.001, Mixed Models Analysis

30. Secondary Outcome: Muscle Strength - Upper Limbs
Description: Muscle strength was evaluated using maximal dynamic strength test [1RM])
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
Kg
  Pre | 21.9 (8.8) | 23.2 (8.4) | 23.2 (8.6)
  Post | 26.9 (10.3) | 28.1 (8.7) | 19.2 (7.5)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p < 0.001, Mixed Models Analysis

31. Secondary Outcome: Muscle Strength - Lower Limbs
Description: Muscle strength was evaluated using maximal dynamic strength test [1RM])
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
Kg
  Pre | 99.9 (35.6) | 99.6 (35.7) | 106.9 (43.0)
  Post | 120.8 (39.7) | 124.8 (36.5) | 94.3 (43.4)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p < 0.001, Mixed Models Analysis

32. Secondary Outcome: Muscle Function (Short Physical Performance Battery)
Description: Muscle function evaluated through battery of tests - Short Physical Performance Battery (SPPB). The SPPB is a standardized assessment of lower extremity function that includes three components: balance tests, gait speed over 4 meters, and the five-times sit-to-stand test. Each component is scored from 0 to 4, with a total score ranging from 0 to 12. Higher scores indicate better physical performance. The SPPB is widely used to evaluate physical function, predict disability, and monitor health status in older adults.
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
score on a scale
  Pre | 8.9 (2.1) | 8.2 (2.2) | 9.3 (1.6)
  Post | 10.7 (1.6) | 10.9 (1.9) | 9.0 (1.6)

33. Secondary Outcome: Muscle Function (30-s Sit-to-stand Test)
Description: The 30-second sit-to-stand test is a simple measure of lower body strength and functional capacity. Participants are asked to rise from a seated position and sit back down as many times as possible within 30 seconds. The total number of complete sit-to-stand repetitions performed in the given time is recorded. This test is commonly used to assess physical fitness and mobility, particularly in older adults or individuals with health conditions.
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: number of repetitions
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
number of repetitions
  Pre | 10.3 (3.5) | 9.4 (3.2) | 10.4 (3.1)
  Post | 12.8 (3.9) | 12.4 (3.5) | 10.2 (2.4)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p < 0.001, Mixed Models Analysis

34. Secondary Outcome: Muscle Function (Timed-up-and-go)
Description: The Timed Up and Go (TUG) test is a simple and widely used assessment of mobility and balance. Participants are asked to stand up from a seated position, walk 3 meters, turn around, walk back to the chair, and sit down again, all as quickly as possible. The total time taken to complete the task is recorded. The TUG test is commonly used to evaluate functional mobility, fall risk, and the ability to perform daily activities, particularly in older adults or individuals with mobility impairments.
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
seconds
  Pre | 9.76 (4.10) | 10.91 (4.26) | 8.67 (1.79)
  Post | 8.49 (2.97) | 9.01 (4.37) | 9.38 (1.84)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p < 0.001, Mixed Models Analysis

35. Secondary Outcome: Muscle Function (Gait Speed)
Description: Muscle function evaluated through 4-m gait speed test. The 4-meter usual gait speed test measures the time it takes for a participant to walk a distance of 4 meters at their usual pace. The test is commonly used to assess walking speed, which is an important indicator of mobility, physical function, and overall health. The time taken to complete the 4-meter walk is recorded and used to evaluate the individual's functional capacity, with slower times potentially indicating mobility impairments or a higher risk of adverse health outcomes.
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
m/s
  Pre | 0.95 (0.23) | 0.90 (0.25) | 0.98 (0.18)
  Post | 1.13 (0.26) | 1.13 (0.27) | 0.97 (0.18)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p < 0.001, Mixed Models Analysis

36. Secondary Outcome: Cardiorespiratory Fitness
Description: Cardiorespiratory fitness was evaluated by maximal oxygen uptake (VO²max) during a maximal exercise test on a treadmill
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: mL/Kg/min
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
mL/Kg/min
  Pre | 16.0 (4.4) | 17.7 (3.2) | 17.6 (3.6)
  Post | 19.2 (5.4) | 20 (2.6) | 17.9 (3.4)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p < 0.001, Mixed Models Analysis

37. Secondary Outcome: Insulin Sensitivity as Assessed by Surrogates of Insulin Sensitivity
Description: Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) is a method used to estimate insulin resistance based on fasting plasma glucose and fasting insulin levels. It is calculated using the following formula:
  HOMA-IR = (fasting insulin [µU/mL] × fasting glucose [mg/dL]) / 405. Higher values of HOMA-IR indicate greater insulin resistance and are considered worse. There is no fixed theoretical maximum value, but typical reference ranges in healthy individuals are usually <2. Values above this threshold may suggest impaired insulin sensitivity or metabolic dysfunction. The HOMA-IR is widely used in clinical and research settings as a surrogate marker for insulin resistance.
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
Index
  Pre | 4.2 (0.2) | 4.3 (0.2) | 4.1 (0.1)
  Post | 2.5 (0.2) | 3.1 (0.2) | 3.6 (0.2)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.017, Mixed Models Analysis

38. Secondary Outcome: Brachial Flow-mediated Dilation (FMD)
Description: Brachial flow-mediated dilation (FMD) is a non-invasive measure of endothelial function, assessed using high-resolution B-mode ultrasound. The test evaluates the percent change in brachial artery diameter in response to increased blood flow (reactive hyperemia) following 3 minutes of cuff occlusion, on the forearm. An increase in arterial diameter after cuff release indicates vasodilation mediated by nitric oxide. Higher FMD values reflect better endothelial function, whereas lower values are associated with cardiovascular risk and impaired vascular health.
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: percentage of flow mediated dilatation
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
percentage of flow mediated dilatation
  Pre | 4.6 (0.5) | 4.8 (0.5) | 5 (0.6)
  Post | 7.8 (0.6) | 6.3 (0.6) | 2.6 (0.6)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p < 0.001, Mixed Models Analysis

39. Other Pre Specified Outcome: Lipid Profile (HDL)
Description: Lipid profile (i.e; HDL, LDL, VLDL, and triglycerides) were evaluated by colorimetric enzymatic methods
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
mg/dL
  Pre | 52.1 (0.9) | 52.8 (0.9) | 52.8 (0.9)
  Post | 51.4 (0.9) | 51.5 (0.9) | 51.7 (0.9)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.949, Mixed Models Analysis

40. Other Pre Specified Outcome: Lipid Profile (LDL)
Description: Lipid profile (i.e; HDL, LDL, VLDL, and triglycerides) were evaluated by colorimetric enzymatic methods
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
mg/dL
  Pre | 116.1 (3.4) | 115.5 (3.5) | 116.8 (3.5)
  Post | 111.1 (3.8) | 111.4 (3.6) | 112.3 (3.7)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.993, Mixed Models Analysis

41. Other Pre Specified Outcome: Lipid Profile (VLDL)
Description: Lipid profile (i.e; HDL, LDL, VLDL, and triglycerides) were evaluated by colorimetric enzymatic methods
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
mg/dL
  Pre | 25.2 (0.7) | 25.4 (0.7) | 25.1 (0.7)
  Post | 22.8 (0.8) | 22.8 (0.8) | 23.9 (0.8)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.601, Mixed Models Analysis

42. Other Pre Specified Outcome: Lipid Profile (Triglycerides)
Description: Lipid profile (i.e; HDL, LDL, VLDL, and triglycerides) were evaluated by colorimetric enzymatic methods
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
mg/dL
  Pre | 140.4 (4.9) | 141.1 (5) | 138.8 (5.1)
  Post | 119.0 (5.3) | 122.5 (5.3) | 130.8 (5.4)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.408, Mixed Models Analysis

43. Other Pre Specified Outcome: Telomere Length
Description: Relative telomere length was measured using quantitative polymerase chain reaction (qPCR), which determines the ratio of telomeric repeat copy number (T) to a single-copy gene number (S) in a given sample. This T/S ratio is a unitless index that reflects the average telomere length relative to the reference gene. Higher T/S ratios indicate longer telomeres, while lower values indicate shorter telomeres. Although the T/S ratio does not provide absolute telomere length in base pairs, it is a widely used, validated method to assess relative telomere length in epidemiological and clinical research.
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Population: This analysis was conducted in a subsample of participants who completed the study protocol. Two participants from the CREX+PTN group and two participants from the CREX+PLA group were excluded from the analysis due to sample quality issues.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 27 | 27 | 27
Ratio
  Pre | 0.98 (0.05) | 0.97 (0.05) | 0.99 (0.05)
  Post | 0.99 (0.06) | 0.99 (0.04) | 0.99 (0.05)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.082, Mixed Models Analysis

44. Other Pre Specified Outcome: Oxidative Stress - Superoxide Dismutase
Description: Superoxide dismutase (SOD) activity was measured using an enzyme-linked immunosorbent assay (ELISA), following the manufacturer's instructions. The assay is based on the competitive binding of SOD present in the sample and a SOD standard to a monoclonal antibody coated on a microplate.
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Population: as for outcome 43
Measure: Mean (Standard Deviation); unit: percentage inhibition per 2 µL of samp
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 27 | 27 | 27
percentage inhibition per 2 µL of samp
  Pre | 22.6 (5.8) | 21.5 (4.0) | 21.5 (5.5)
  Post | 23.2 (4.9) | 23.3 (4.1) | 22.6 (4.5)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.550, Mixed Models Analysis

45. Other Pre Specified Outcome: Oxidative Stress - Catalase Activity
Description: Catalase activity was assessed using an enzyme-linked immunosorbent assay (ELISA), according to the manufacturer's protocol. The assay quantifies catalase based on the competition between the sample catalase and a catalase standard for binding to specific antibodies coated on the microplate. The detection is achieved through a colorimetric reaction measured at a specific wavelength.
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Population: as for outcome 43
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 27 | 27 | 27
U/mL
  Pre | 6.2 (2.3) | 6.6 (0.8) | 5.8 (2.7)
  Post | 6.0 (2.6) | 6.8 (0.8) | 5.7 (2.3)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.700, Mixed Models Analysis

46. Other Pre Specified Outcome: Oxidative Stress - Glutathione Peroxidase
Description: Glutathione peroxidase activity was measured using a colorimetric assay according to the manufacturer's instructions. The method is based on the enzyme-catalyzed reduction of hydrogen peroxide by reduced glutathione (GSH), forming oxidized glutathione (GSSG). In the presence of glutathione reductase and NADPH, GSSG is converted back to GSH with concomitant oxidation of NADPH to NADP⁺.
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Population: as for outcome 43
Measure: Mean (Standard Deviation); unit: µmol GSH/min/mL
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 27 | 27 | 27
µmol GSH/min/mL
  Pre | 404.2 (52.8) | 406.5 (49.5) | 401.2 (40.7)
  Post | 416.3 (45.7) | 412.5 (47.9) | 396.1 (39.0)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.254, Mixed Models Analysis

47. Other Pre Specified Outcome: Oxidative Stress - Glutathione Reductase
Description: Oxidative stress markers (SOD, CAT, glutathione, GPx, GST and TBARS) were assessed through ELISA assay.
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Population: as for outcome 43
Measure: Mean (Standard Deviation); unit: µmol NADPH/min/mL
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 27 | 27 | 27
µmol NADPH/min/mL
  Pre | 48.7 (3.2) | 48.0 (3.0) | 48.4 (2.4)
  Post | 49.6 (4.2) | 47.3 (4.8) | 49.1 (2.5)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.373, Mixed Models Analysis

48. Other Pre Specified Outcome: Oxidative Stress - Glutathione S-transferases
Description: Glutathione S-transferase (GST) activity was assessed using a colorimetric assay based on the conjugation of the substrate 1-chloro-2,4-dinitrobenzene (CDNB) with reduced glutathione (GSH). The reaction results in a yellow product that is quantified by measuring the absorbance at 340 nm.
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Population: as for outcome 43
Measure: Mean (Standard Deviation); unit: pmol GSH conjugates/min/mL
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 27 | 27 | 27
pmol GSH conjugates/min/mL
  Pre | 17.4 (6.5) | 18.7 (11.6) | 18.3 (9.3)
  Post | 21.3 (7.1) | 19.8 (9.6) | 18.6 (9.2)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.407, Mixed Models Analysis

49. Other Pre Specified Outcome: Oxidative Stress - Thiobarbituric Acid Reactive Substances
Description: Thiobarbituric Acid Reactive Substances (TBARS): Lipid peroxidation was assessed by measuring thiobarbituric acid reactive substances (TBARS), following the manufacturer's instructions. This colorimetric assay detects malondialdehyde (MDA), a byproduct of lipid peroxidation, which reacts with thiobarbituric acid to form a colored complex measurable at 532-535 nm. Results are expressed as micromoles of MDA equivalents per liter (µmol/L), with higher values indicating greater oxidative stress.
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Population: as for outcome 43
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 27 | 27 | 27
µmol/L
  Pre | 2.05 (0.93) | 2.06 (1.20) | 1.94 (0.52)
  Post | 1.97 (0.84) | 2.15 (1.21) | 2.25 (0.97)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.051, Mixed Models Analysis

50. Other Pre Specified Outcome: Inflammatory Profile - IL1β
Description: Inflammatory profile (i.e.; IL1β, IL-10, IL-6, and TNF-α) were quantified using the Luminex xMAP technology.
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
pg/mL
  Pre | 1.45 (0.37) | 1.33 (0.37) | 1.01 (0.38)
  Post | 1.46 (0.37) | 0.88 (0.37) | 1.22 (0.38)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.385, Mixed Models Analysis

51. Other Pre Specified Outcome: Inflammatory Profile - IL-10
Description: Inflammatory profile (i.e.; IL1β, IL-10, IL-6, and TNF-α) were quantified using the Luminex xMAP technology.
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
pg/mL
  Pre | 3.75 (0.75) | 4.46 (0.76) | 3.56 (0.77)
  Post | 3.78 (0.75) | 2.47 (0.76) | 3.96 (0.77)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.239, Mixed Models Analysis

52. Other Pre Specified Outcome: Inflammatory Profile - IL-6
Description: Inflammatory profile (i.e.; IL1β, IL-10, IL-6, and TNF-α) were quantified using the Luminex xMAP technology.
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
pg/mL
  Pre | 3.30 (0.46) | 2.99 (0.46) | 2.92 (0.47)
  Post | 2.49 (0.46) | 2.49 (0.46) | 3.25 (0.47)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.463, Mixed Models Analysis

53. Other Pre Specified Outcome: Inflammatory Profile - TNF-α
Description: Inflammatory profile (i.e.; IL1β, IL-10, IL-6, and TNF-α) were quantified using the Luminex xMAP technology.
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
pg/mL
  Pre | 20.1 (1.2) | 19.6 (1.2) | 19.4 (1.2)
  Post | 14.7 (1.2) | 15.5 (1.2) | 20.1 (1.2)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.032, Mixed Models Analysis

54. Other Pre Specified Outcome: Inflammatory Profile - C-Reactive Protein
Description: Inflammatory profile (i.e.; C-Reactive Protein ) was quantified via an immunoturbidimetric assay.
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
pg/mL
  Pre | 5.76 (0.79) | 5.19 (0.81) | 6.01 (0.83)
  Post | 4.25 (0.87) | 5.74 (0.86) | 5.54 (0.87)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.469, Mixed Models Analysis

55. Other Pre Specified Outcome: Area Under the Curve (AUC) of Blood Glucose
Description: The area under the curve (AUC) of blood glucose was measured during a 2-hour oral glucose tolerance test (OGTT). Blood samples were collected at baseline (0 minutes, following a 12-hour overnight fast), and at 30, 60, 90, and 120 minutes after ingestion of a 75 g glucose bolus. The AUC was calculated using these time points (0, 30, 60, 90, and 120 minutes) to assess the blood glucose response over the 2-hour period following glucose ingestion.
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (95% Confidence Interval); unit: mg·min/dL
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
mg·min/dL
  Pre | 683.54 [617.38 to 749.70] | 641.73 [574.51 to 708.94] | 648.99 [581.77 to 716.20]
  Post | 599.51 [533.35 to 665.66] | 622.22 [555.00 to 689.43] | 638.20 [570.98 to 705.41]
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.013, Mixed Models Analysis

56. Other Pre Specified Outcome: Area Under the Curve (AUC) of Insulin
Description: The area under the curve (AUC) of insulin was measured during a 2-hour oral glucose tolerance test (OGTT). Blood samples were collected at baseline (0 minutes, following a 12-hour overnight fast), and at 30, 60, 90, and 120 minutes after ingestion of a 75 g glucose bolus. The AUC was calculated using these time points (0, 30, 60, 90, and 120 minutes) to assess the insulin response over the 2-hour period following glucose ingestion.
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (95% Confidence Interval); unit: μU·min/mL
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
μU·min/mL
  Pre | 442.08 [355.59 to 528.58] | 417.23 [329.35 to 505.11] | 432.69 [344.81 to 520.57]
  Post | 259.90 [173.40 to 346.39] | 310.21 [222.34 to 398.09] | 403.40 [315.52 to 491.28]
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.064, Mixed Models Analysis

57. Other Pre Specified Outcome: Anxiety
Description: Anxiety was assessed using the Geriatric Anxiety Inventory (GAI), a 20-item self-report questionnaire designed to measure anxiety symptoms in older adults. The total score ranges from 0 to 20, with higher scores reflecting more severe anxiety symptoms.
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
score on a scale
  Pre | 6.8 (5.0) | 6.6 (4.8) | 4.4 (3.8)
  Post | 4.6 (5.1) | 5.5 (5.3) | 4.0 (4.1)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.0314, Mixed Models Analysis

58. Other Pre Specified Outcome: Depression
Description: Depression was assessed using the Geriatric Depression Scale (GDS-15), a 15-item self-report questionnaire designed to measure depressive symptoms in older adults. The total score ranges from 0 to 15, with higher scores indicating more severe depression.
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
score on a scale
  Pre | 4.1 (2.9) | 4.8 (3.4) | 2.8 (4.4)
  Post | 2.6 (2.8) | 2.6 (2.8) | 2.5 (4.0)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.0147, Mixed Models Analysis

59. Other Pre Specified Outcome: Health-related Quality of Life - Physical Component
Description: Health-related quality of life was evaluated using the 36-Item Short Form Health Survey (SF-36), a widely used questionnaire designed to assess various dimensions of health in adults. The total score ranges from 0 to 100, with higher scores indicating better health-related quality of life.
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
score on a scale
  Pre | 61.2 (24.3) | 63.9 (22.1) | 71.8 (19.7)
  Post | 77.2 (19.8) | 77.2 (19.5) | 75.6 (18.3)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.007, Mixed Models Analysis

60. Other Pre Specified Outcome: Health-related Quality of Life - Mental Component
Description: as for outcome 59
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
score on a scale
  Pre | 59.3 (22.4) | 58.9 (23.3) | 63.0 (19.0)
  Post | 74.8 (17.3) | 81.5 (13.4) | 64.5 (21.1)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p < 0.001, Mixed Models Analysis

61. Other Pre Specified Outcome: Sleep Quality
Description: Sleep quality was assessed using the Pittsburgh Sleep Quality Index (PSQI), a self-report questionnaire that evaluates various aspects of sleep quality. The PSQI is scored by summing the scores of seven components, each ranging from 0 to 3. The total score ranges from 0 to 21, with higher scores indicating poorer sleep quality.
Time Frame: Baseline (Pre-intervention) and 16 weeks (Post-intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
Number analyzed (Participants) | 35 | 35 | 35
score on a scale
  Pre | 5.9 (3.2) | 7.2 (3.6) | 5.6 (3.0)
  Post | 4.6 (3.1) | 3.6 (2.1) | 5.0 (3.7)
Statistical Analysis 1: Comparison: Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) vs Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) vs Control Group (CTRL); Test type: Superiority; p = 0.001, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) | Control Group (CTRL)
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 1/35 | 1/35 | 0/35
Other Adverse Events (participants affected / at risk) | 8/35 | 8/35 | 8/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) (N=35) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) (N=35) | Control Group (CTRL) (N=35)
Third-degree atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Caloric Restriction Associated to Exercise Training Plus Protein Supplementation (CREX+PTN) (N=35) | Caloric Restriction Associated to Exercise Training Plus Isocaloric Placebo (CREX+PLA) (N=35) | Control Group (CTRL) (N=35)
Articular pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Fell during exercise training (General disorders) | 1 (1) | 0 (0) | 0 (0)
Transitory pain after muscle biopsies (Musculoskeletal and connective tissue disorders) | 6/6 (6) | 6/7 (6) | 6/7 (6)
Bruising after muscle biopsies (Musculoskeletal and connective tissue disorders) | 0/6 (0) | 1/7 (1) | 1/7 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-23): https://cdn.clinicaltrials.gov/large-docs/66/NCT04981366/Prot_SAP_000.pdf